CLINICAL TRIAL: NCT06407934
Title: A Phase 3, Multinational, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel Group 52-week Extension Study to Evaluate the Treatment Response and Safety of Two Amlitelimab Dose Regimens Administered by Subcutaneous Injection in Participants Aged 12 Years and Older With Moderate-to-severe Atopic Dermatitis
Brief Title: A Study to Evaluate the Treatment Response and Safety of Two Dose Regimens of Subcutaneous Amlitelimab Compared With Treatment Withdrawal in Participants Aged 12 Years and Older With Moderate-to-severe Atopic Dermatitis
Acronym: ESTUARY
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC17600; U1111-1290-9215 (Registry Identifier: ICTRP); 2023-508096-36 (Registry Identifier: CTIS)
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Dermatitis Atopic
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Amlitelimab dose 1 (Experimental): Subcutaneous injection as per protocol
  Interventions: Drug: Amlitelimab
- Amlitelimab dose 2 (Experimental): Subcutaneous injection as per protocol
  Interventions: Drug: Amlitelimab
- Placebo (Placebo Comparator): Subcutaneous injection as per protocol
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amlitelimab — Pharmaceutical form: Injection solution
  Route of administration: Subcutaneous (SC) injection
  Other Names: SAR445229
  Arms: Amlitelimab dose 1; Amlitelimab dose 2
Drug: Placebo — Pharmaceutical form: Injection solution
  Route of administration: SC injection
  Arms: Placebo

SUMMARY:
This is a multinational, multicenter, randomized, double-blind, placebo-controlled, parallel, Phase 3 study for treatment of participants aged 12 years and older diagnosed with moderate-to-severe atopic dermatitis (AD).

The main objective of this study is to evaluate if those participants who received amlitelimab dose 1 in the parent studies (EFC17559 [COAST-1], EFC17560 [COAST 2], EFC17561 [SHORE]) and were responders can maintain their response either remaining at dose 1 or switching to dose 2 of amlitelimab compared to treatment withdrawal.

Study details include:

The study duration will be up to 68 weeks including a 52-week randomized double-blind period, and a 16-week safety follow-up for participants not entering the LTS17367 (RIVER-AD).

The study duration will be up to 52 weeks for participants entering the LTS17367 [RIVER-AD] study at the Week 52 visit of EFC17600 (ESTUARY).

The total treatment duration will be up to 52 weeks. The total number of visits will be up to 15 visits (or 14 visits for those entering LTS17367 [RIVER-AD] study).

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at least 12 years of age inclusive, at the time the informed consent is signed.
* Must have participated, received study treatment without permanent investigational medicinal product (IMP) discontinuation, and adequately completed the assessments required for the treatment period in one of the three 24-week parent studies EFC17559 (COAST-1), EFC17560 (COAST-2) or EFC17561 (SHORE) for moderate-to-severe AD.
* Able and willing to comply with requested study visit and procedures.
* Body weight must be ≥ 25 kg.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Developed a medical condition that would preclude participation as described in Exclusion Criteria or Permanent Discontinuation of EFC17559 (COAST-1)/EFC17560 (COAST-2)/EFC17561 (SHORE) clinical trial protocols.
* Having received any prohibited medication or procedure for AD that resulted in IMP discontinuation in the parent study EFC17559 (COAST-1), EFC17560 (COAST-2) or EFC17561 (SHORE).
* Participants who, during their participation in the parent study EFC17559 (COAST-1) /EFC17560 (COAST-2)/EFC17561 (SHORE), developed an adverse event (AE) or a serious adverse event (SAE) deemed related to amlitelimab, which in the opinion of the Investigator could indicate that continued treatment with amlitelimab may present an unreasonable risk for the participant.
* Participants who have had IMP permanently discontinued for any reason before or at the time of the planned first dose in the EFC17600 (ESTUARY) study.
* Conditions in the parent study EFC17559 (COAST-1)/EFC17560 (COAST-2)/EFC17561 (SHORE) that led to Investigator - or Sponsor-initiated withdrawal of participant from the study (eg, non-compliance, inability to complete study assessments, etc.).
* Participant not suitable for participation, whatever the reason, as judged by the Investigator, including medical or clinical conditions, or participants potentially at risk of noncompliance to study procedures.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1541 (Actual)
Dates: Start 2024-05-08 (Actual); Primary Completion 2026-06-29 (Estimated); Study Completion 2027-03-17 (Estimated)

PRIMARY OUTCOMES:
Responders from parent studies: Proportion of participants who maintain treatment response in ESTUARY. | Week 48
  Maintenance of clinical response is defined as having validated Investigator Global Assessment scale for atopic dermatitis (vIGA-AD) 0 (clear) or 1 (almost clear) OR 75% reduction in Eczema Area and Severity Index (EASI) compared to parent study baseline EASI (EASI-75^) OR vIGA-AD 0 (clear) or 1 (almost clear) and EASI-75^.
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD.

SECONDARY OUTCOMES:
Responders from parent studies: Proportion of participants who continue to be EASI-75^ among the participants who met EASI-75^ at baseline of ESTUARY | Up to Week 48
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD. EASI-75 is 75% reduction from baseline in EASI score. The symbol ^ represents "based on parent study baseline".
Responders from parent studies: Proportion of participants who continue to be vIGA-AD 0 (clear) or 1 (almost clear) among participants who met vIGA-AD 0 (clear) or 1 (almost clear) at baseline of ESTUARY | Up to Week 48
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).
Responders from parent studies: Proportion of participants who continue to be vIGA-AD 0 or 1 with presence of only barely perceptible erythema among those who are vIGA-AD 0 or 1 with presence of only barely perceptible erythema at baseline of ESTUARY | Up to Week 48
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear), 1 (almost clear) to 4 (severe). Barely perceptible erythema with no induration/papulation, no lichenification, no oozing or crusting.
Responders from parent studies: Proportion of participants who maintained weekly average of daily PP-NRS reduction of ≥4^ among the participants with weekly average of daily PP-NRS reduction of ≥4^ at baseline of ESTUARY | Up to Week 48
  The Peak Pruritus-Numerical Rating Scale (PP-NRS) is a validated single item 0-10 numeric rating scale assessing peak pruritus (itch) associated with AD with 0 = no itch and 10 = worst itch imaginable. The symbol ^ represents "based on parent study baseline".
Responders from parent studies: Proportion of participants who maintain vIGA-AD ≤1 and PP-NRS ≤1 at Week 48 of ESTUARY among participants who were vIGA-AD ≤1 and PP-NRS ≤1 at baseline of ESTUARY | Up to Week 48
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe). The PP-NRS is a validated single item 0-10 numeric rating scale assessing peak pruritus (itch) associated with AD with 0 = no itch and 10 = worst itch imaginable.
Responders from parent studies: Proportion of participants who maintain vIGA-AD ≤2 and PP-NRS ≤4 at Week 48 of ESTUARY among participants who were vIGA-AD ≤2 and PP-NRS ≤4 at baseline of ESTUARY | Up to Week 48
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe). The PP-NRS is a validated single item 0-10 numeric rating scale assessing peak pruritus (itch) associated with AD with 0 = no itch and 10 = worst itch imaginable.
Responders from parent studies: Proportion of participants who maintain treatment response | Up to Week 44
  Maintenance of treatment response is defined as having vIGA-AD 0 (clear) or 1 (almost clear) OR 75% reduction in EASI compared to parent study baseline EASI (EASI-75^) OR vIGA-AD 0 (clear) or 1 (almost clear) and EASI-75^. The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD.
Responders from parent studies: Percent change in EASI from parent study baseline | Parent study baseline to Week 48
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD.
Responders from parent studies: Proportion of participants who maintained EASI-75^ among the participants who met EASI-75^ at baseline of ESTUARY | Up to Week 48
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD. EASI-75^ is 75% reduction from baseline in EASI score. The symbol ^ represents "based on parent study baseline".
Responders from parent studies: Proportion of participants with EASI-75^ | Parent study baseline to Week 48
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD. EASI-75 is 75% reduction from baseline in EASI score. The symbol ^ represents "based on parent study baseline".
Responders from parent studies: Proportion of participants who continue to be EASI-50^ among the participants who met EASI-50^ at baseline of ESTUARY | Up to Week 48
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD. EASI-50 is 50% reduction from baseline in EASI score. The symbol ^ represents "based on parent study baseline".
Responders from parent studies: Proportion of participants with EASI-50^ | Parent study baseline to Week 48
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD. EASI-50 is 50% reduction from baseline in EASI score. The symbol ^ represents "based on parent study baseline".
Responders from parent studies: Proportion of participants who continue to be EASI-90^ among the participants who met EASI-90^ at baseline of ESTUARY | Up to Week 48
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD. EASI-90 is 90% reduction from baseline in EASI score. The symbol ^ represents "based on parent study baseline".
Responders from parent studies: Proportion of participants with EASI-90^ | Parent study baseline to Week 48
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD. EASI-90 is 90% reduction from baseline in EASI score. The symbol ^ represents "based on parent study baseline".
Responders from parent studies: Proportion of participants who continue to be EASI-100^ among the participants who met EASI-100^ at baseline of ESTUARY | Up to Week 48
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD. EASI-100 is 100% reduction from baseline in EASI score. The symbol ^ represents "based on parent study baseline".
Responders from parent studies: Proportion of participants with EASI-100^ | Parent study baseline to Week 48
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD. EASI-100 is 100% reduction from baseline in EASI score. The symbol ^ represents "based on parent study baseline".
Responders from parent studies: Time to the first event of loss of EASI-75^ response among the participants who were EASI-75^ responders at baseline of ESTUARY | Up to Week 48
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD. EASI-75 is 75% reduction from baseline in EASI score. The symbol ^ represents "based on parent study baseline".
Responders from parent studies: Time to the first event of loss of EASI-50^ response among the participants who were EASI-50^ responders at baseline of ESTUARY | Up to Week 48
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD. EASI-50 is 50% reduction from baseline in EASI score. The symbol ^ represents "based on parent study baseline".
Responders from parent studies: Time to the first event of loss of EASI-90^ response among the participants who were EASI-90^ responders at baseline of ESTUARY | Up to Week 48
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD. EASI-90 is 90% reduction from baseline in EASI score. The symbol ^ represents "based on parent study baseline".
Responders from parent studies: Time to the first event of loss of EASI-100^ among participants who were EASI-100^ at baseline of ESTUARY | Up to Week 48
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD. EASI-100^ is 100% reduction from baseline in EASI score. The symbol ^ represents "based on parent study baseline".
Responders from parent studies: Proportion of participants with vIGA-AD 0 (clear) or 1 (almost clear) | Up to Week 48
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).
Responders from parent studies: Proportion of participants who are vIGA-AD 0 (clear) or 1 (almost clear) with presence of only barely perceptible erythema (no induration/papulation, no lichenification, no oozing or crusting) | Up to Week 48
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).
Responders from parent studies: Time to first event of vIGA-AD ≥1 among those participants who were vIGA-AD 0 (clear) at baseline of ESTUARY | Up to Week 48
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).
Responders from parent studies: Time to first event of vIGA-AD ≥2 among those participants who were vIGA AD 0 (clear) or 1 (almost clear) at baseline of ESTUARY | Up to Week 48
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).
Responders from parent studies: Time to first event of vIGA-AD ≥3 (moderate or severe) among those participants who were vIGA-AD 0 (clear) or 1 (almost clear) at baseline of ESTUARY | Up to Week 48
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).
Responders from parent studies: Time to first event of vIGA-AD ≥3 (moderate or severe) among those participants who were vIGA-AD 0 (clear) at baseline of ESTUARY | Up to Week 48
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).
Responders from parent studies: Proportion of participants who have an increase of ≥2 points in vIGA-AD from ESTUARY baseline among the participants who were vIGA-AD 0 (clear) or 1 (almost clear) at baseline of ESTUARY | Up to Week 48
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).
Responders from parent studies: Proportion of participants who have an increase of ≥2 points in vIGA-AD from ESTUARY baseline among the participants who were vIGA-AD 3 (moderate) at baseline of parent study | Up to Week 48
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).
Responders from parent studies: Proportion of participants who have an increase of ≥2 points in vIGA-AD from ESTUARY baseline among the participants who were vIGA-AD 4 (severe) at baseline of parent study | Up to Week 48
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).
Responders from parent studies: Proportion of participants with vIGA-AD 0 (clear) or 1 (almost clear) and/or EASI-75^ among the participants who were vIGA-AD 0 (clear) or 1 (almost clear) and/or EASI-75^ at baseline of ESTUARY | Up to Week 48
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe). The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD. EASI-75 is 75% reduction from baseline in EASI score. The symbol ^ represents "based on parent study baseline".
Responders from parent studies: Proportion of participants with ≥ 4 points reduction in weekly average of daily PP-NRS from parent study baseline | Parent study baseline to Week 48
  The PP-NRS is a validated single item 0-10 numeric rating scale assessing peak pruritus (itch) associated with AD with 0 = no itch and 10 = worst itch imaginable.
Responders from parent studies: Percent change in weekly average of daily PP-NRS from parent study baseline | Parent study baseline to Week 48
  The PP-NRS is a validated single item 0-10 numeric rating scale assessing peak pruritus (itch) associated with AD with 0 = no itch and 10 = worst itch imaginable.
Responders from parent studies: Absolute change in weekly average of daily PP-NRS from parent study baseline | Parent study baseline to Week 48
  The PP-NRS is a validated single item 0-10 numeric rating scale assessing peak pruritus (itch) associated with AD with 0 = no itch and 10 = worst itch imaginable.
Responders from parent studies: Proportion of participants who maintained PP-NRS 0 or 1 among the participants who were PP-NRS 0 or 1 at baseline of ESTUARY | Up to Week 48
  The PP-NRS is a validated single item 0-10 numeric rating scale assessing peak pruritus (itch) associated with AD with 0 = no itch and 10 = worst itch imaginable.
Responders from parent studies:Proportion of participants who maintained vIGA-AD 0 or 1 and/or EASI-75^ and weekly average of daily (WAD) PP-NRS reduction ≥4^ among those who were vIGA-AD 0 or 1 and/or EASI-75^ and WAD PP-NRS reduction ≥4^ at ESTUARY BL | Up to Week 48
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear), 1 (almost clear) to 4 (severe). The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD. EASI-75 is 75% reduction from baseline in EASI score. The Peak Pruritus-Numerical Rating Scale (PP-NRS) is a validated single item 0-10 numeric rating scale assessing peak pruritus (itch) associated with AD with 0 = no itch and 10 = worst itch imaginable. The symbol ^ represents "based on parent study baseline". BL=baseline.
Responders from parent studies: Proportion of participants who continue to be vIGA-AD 0 (clear) among the participants who were vIGA- AD 0 (clear) at baseline of ESTUARY | Up to Week 48
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).
Responders from parent studies: Proportion of participants who maintain vIGA-AD 0 to 2 (clear, almost clear, and mild disease) among participants who were vIGA-AD 0 to 2 (clear, almost clear, and mild disease) at baseline of ESTUARY | Up to Week 48
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).
Responders from parent studies: Proportion of participants who maintain PP-NRS ≤4 among participants who were PP-NRS ≤4 at baseline of ESTUARY | Up to Week 48
  The PP-NRS is a validated single item 0-10 numeric rating scale assessing peak pruritus (itch) associated with AD with 0 = no itch and 10 = worst itch imaginable.
Responders from parent studies: Absolute change in weekly average of daily SD-NRS from parent study baseline | Parent study baseline to Week 48
  The Sleep Disturbance-Numerical Rating Scale (SD-NRS) is a single item 0-10 numeric rating scale assessing sleep disturbance associated with AD with 0 = no sleep loss and 10 = did not sleep at all.
Responders from parent studies: Proportion of participants who maintained weekly average of daily SD-NRS reduction of ≥3^ among the participants with weekly average of daily SD-NRS reduction of ≥3^ at baseline of ESTUARY | Up to Week 48
  The SD-NRS is a single item 0-10 numeric rating scale assessing sleep disturbance associated with AD with 0 = no sleep loss and 10 = did not sleep at all. The symbol ^ represents "based on parent study baseline".
Responders from parent studies: Proportion of participants with ≥3 points reduction in weekly average of daily SD-NRS from parent study baseline | Parent study baseline to Week 48
  The SD-NRS is a single item 0-10 numeric rating scale assessing sleep disturbance associated with AD with 0 = no sleep loss and 10 = did not sleep at all.
Responders from parent studies: Proportion of participants with ≥4 points reduction in weekly average of daily SP-NRS from parent study baseline | Parent study baseline to Week 48
  The Skin Pain-Numerical Rating Scale (SP-NRS) is a single item 0-10 numeric rating scale assessing skin pain associated with AD with 0 = no pain and 10 = worst possible pain imaginable.
Responders from parent studies: Proportion of participants who maintained weekly average of daily SP-NRS reduction of ≥4^ among the participants with weekly average of daily SP-NRS reduction of ≥4^ at ESTUARY baseline | Up to Week 48
  The SP-NRS is a single item 0-10 numeric rating scale assessing skin pain associated with AD with 0 = no pain and 10 = worst possible pain imaginable. The symbol ^ represents "based on parent study baseline".
Responders from parent studies: Absolute change in weekly average of daily SP-NRS from parent study baseline | Parent study baseline to Week 48
  The SP-NRS is a single item 0-10 numeric rating scale assessing skin pain associated with AD with 0 = no pain and 10 = worst possible pain imaginable.
Responders from parent studies: Proportion of participants who maintained SCORAD ≥8.7^ among participants with reduction in SCORAD ≥8.7^ at baseline of ESTUARY | Up to Week 48
  The Scoring Atopic Dermatitis (SCORAD) index is a clinical tool to evaluate the extent and severity of AD. Total score ranges from 0 (absent disease) to 103 (severe disease). The symbol ^ represents "based on parent study baseline".
Responders from parent studies: Percent change in SCORAD index from parent study baseline | Parent study baseline to Week 48
  The SCORAD index is a clinical tool to evaluate the extent and severity of AD. Total score ranges from 0 (absent disease) to 103 (severe disease).
Responders from parent studies: Absolute change in SCORAD index from parent study baseline | Parent study baseline to Week 48
  The SCORAD index is a clinical tool to evaluate the extent and severity of AD. Total score ranges from 0 (absent disease) to 103 (severe disease).
Responders from parent studies: Change in percent Body Surface Area (BSA) affected by AD from parent study baseline | Parent study baseline to Week 48
Responders from parent studies: Proportion of participants who maintained POEM ≥4 among the participants with reduction in POEM ≥4 at baseline of ESTUARY | Up to Week 48
  The Patient Oriented Eczema Measure (POEM) is a 7-item self-assessment questionnaire that assesses disease symptoms on a 5-point scale; 0 (no days) to 4 (every day in the last week). The sum of the 7 items gives the total POEM score of 0 (absent disease) to 28 (very severe). Higher scores indicated more severe disease and poor quality of life.
Responders from parent studies: Change in POEM from parent study baseline | Parent study baseline to Week 48
  The POEM is a 7-item self-assessment questionnaire that assesses disease symptoms on a 5-point scale; 0 (no days) to 4 (every day in the last week). The sum of the 7 items gives the total POEM score of 0 (absent disease) to 28 (very severe). Higher scores indicated more severe disease and poor quality of life.
Responders from parent studies: Proportion of participants with a reduction in CDLQI ≥6^ among participants aged ≥12 to <16 years old and with CDLQI baseline ≥6 | Parent study baseline to Week 48
  The Children's Dermatology Quality of Life Index (CDLQI) is a validated 10-item questionnaire to measure dermatology-specific quality of life (QoL) in children aged 4-<16 years. Overall scoring ranges from 0 to 30, with a higher score indicating a poorer QoL. The symbol ^ represents "based on parent study baseline".
Responders from parent studies: Change in CDLQI^ in participants with age ≥12 to <16 years old | Parent study baseline to Week 48
  The CDLQI is a validated 10-item questionnaire to measure dermatology-specific quality of life (QoL) in children aged 4-<16 years. Overall scoring ranges from 0 to 30, with a higher score indicating a poorer QoL. The symbol ^ represents "based on parent study baseline".
Responders from parent studies: Change in Dermatology Life Quality Index (DLQI^) in participants with age ≥16 years among the participants with DLQI ≥4 at parent study baseline | Parent study baseline to Week 48
  The DLQI is a validated 10-item questionnaire to measure dermatology-specific quality of life (QoL) in adult patients. Overall scoring ranges from 0 to 30, with a higher score indicating a poorer QoL. The symbol ^ represents "based on parent study baseline".
Responders from parent studies: Proportion of participants with ≥4 points reduction in DLQI from parent study baseline among the participants with DLQI ≥4 at parent study baseline | Parent study baseline to Week 48
  The DLQI is a validated 10-item questionnaire to measure dermatology-specific quality of life (QoL) in adult patients. Overall scoring ranges from 0 to 30, with a higher score indicating a poorer QoL.
Responders from parent studies: Proportion of participants with HADS-D <8 among the participants who had HADS-D ≥8 at parent study baseline | Parent study baseline to Week 48
  The Hospital Anxiety Depression Scale-Depression (HADS-D) ranges 0-21 with higher score indicating a poorer state.
Responders from parent studies: Proportion of participants with HADS-A <8 among the participants who had HADS-A ≥8 at parent study baseline | Parent study baseline to Week 48
  The Hospital Anxiety Depression Scale-Anxiety (HADS-A) ranges 0-21 with higher score indicating a poorer state.
Responders from parent studies: Proportion of participants requiring rescue medication during the study up to Week 48 of ESTUARY | Up to Week 48
Responders from parent studies: Time to first rescue medication initiation | Up to Week 48
Responders from parent studies: Proportion of participants who are vIGA-AD ≤1 and PP-NRS ≤1 | Up to Week 48
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).
  The PP-NRS is a validated single item 0-10 numeric rating scale assessing peak pruritus (itch) associated with AD with 0 = no itch and 10 = worst itch imaginable.
Responders from parent studies: Proportion of participants who are vIGA-AD ≤2 and PP-NRS ≤4 | Up to Week 48
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).
  The PP-NRS is a validated single item 0-10 numeric rating scale assessing peak pruritus (itch) associated with AD with 0 = no itch and 10 = worst itch imaginable.
Responders from parent studies: Proportion of participants who are "vIGA-AD ≤1 or EASI ≤3" and PP-NRS ≤1 | Up to Week 48
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD.
  The PP-NRS is a validated single item 0-10 numeric rating scale assessing peak pruritus (itch) associated with AD with 0 = no itch and 10 = worst itch imaginable.
Responders from parent studies: Proportion of participants who are "vIGA-AD ≤ 2 or EASI ≤7" AND PP-NRS ≤4 | Up to Week 48
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD.
  The PP-NRS is a validated single item 0-10 numeric rating scale assessing peak pruritus (itch) associated with AD with 0 = no itch and 10 = worst itch imaginable.
Responders from parent studies: Proportion of participants who maintain "vIGA-AD ≤1 or EASI ≤3" AND PP-NRS ≤1 among participants who were "vIGA-AD ≤1 or EASI ≤3" and PP-NRS ≤1 (VLDA) at baseline of ESTUARY | Up to Week 48
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD.
  The PP-NRS is a validated single item 0-10 numeric rating scale assessing peak pruritus (itch) associated with AD with 0 = no itch and 10 = worst itch imaginable.
Responders from parent studies: Proportion of participants who maintain "vIGA-AD ≤2 or EASI ≤7" AND PP-NRS ≤4 among participants who were "vIGA-AD ≤2 or EASI ≤7" AND PP-NRS ≤4 (LDA) at baseline of ESTUARY | Up to Week 48
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD.
  The PP-NRS is a validated single item 0-10 numeric rating scale assessing peak pruritus (itch) associated with AD with 0 = no itch and 10 = worst itch imaginable.
Responders from parent studies: Proportion of participants who are flare free over the 48-week period | Up to Week 48
  Flare is defined as exacerbation of pruritus, assessed using the Peak-Pruritus Numerical Rating Scale (PP-NRS)
Responders from parent studies: For those participants who experience flare, time to first flare | Up to Week 48
  Flare is defined as exacerbation of pruritus, assessed using the Peak-Pruritus Numerical Rating Scale (PP-NRS)
Non-responders from parent studies: Percent change in EASI from parent study baseline | Parent study baseline to Week 48
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD.
Non-responders from parent studies: Proportion of participants with EASI-75^ | Parent study baseline to Week 48
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD. EASI-75 is 75% reduction from baseline in EASI score. The symbol ^ represents "based on parent study baseline".
Non-responders from parent studies: Proportion of participants who continue to be EASI-50^ among the participants who met EASI-50^ at baseline of ESTUARY | Up to Week 48
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD. EASI-50 is 50% reduction from baseline in EASI score. The symbol ^ represents "based on parent study baseline".
Non-responders from parent studies: Proportion of participants with EASI-50^ | Parent study baseline to Week 48
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD. EASI-50 is 50% reduction from baseline in EASI score. The symbol ^ represents "based on parent study baseline".
Non-responders from parent studies: Proportion of participants with EASI-90^ | Parent study baseline to Week 48
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD. EASI-90 is 90% reduction from baseline in EASI score. The symbol ^ represents "based on parent study baseline".
Non-responders from parent studies: Proportion of participants with EASI-100^ | Parent study baseline to Week 48
  The EASI is an Investigator-assessed validated tool used to measure the extent (area) and severity of AD. Total score ranges from 0 to 72 with a higher score indicating increased extent and severity of AD. EASI-100 is 100% reduction from baseline in EASI score. The symbol ^ represents "based on parent study baseline".
Non-responders from parent studies: Proportion of participants with vIGA-AD 0 (clear) or 1 (almost clear) | Up to Week 48
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).
Non-responders from parent studies: Proportion of participants who are vIGA-AD 0 (clear) or 1 (almost clear) with presence of only barely perceptible erythema (no induration/papulation, no lichenification, no oozing or crusting) | Up to Week 48
  The vIGA-AD is an Investigator-completed assessment scale used to determine severity of AD and clinical response to treatment. It is based on a 5-point scale, ranging from 0 (clear) to 4 (severe).
Non-responders from parent studies: Proportion of participants with ≥ 4 points reduction in weekly average of daily PP-NRS from parent study baseline | Parent study baseline to Week 48
  The PP-NRS is a validated single item 0-10 numeric rating scale assessing peak pruritus (itch) associated with AD with 0 = no itch and 10 = worst itch imaginable.
Non-responders from parent studies: Percent change in weekly average of daily PP-NRS from parent study baseline | Parent study baseline to Week 48
  The PP-NRS is a validated single item 0-10 numeric rating scale assessing peak pruritus (itch) associated with AD with 0 = no itch and 10 = worst itch imaginable.
Non-responders from parent studies: Absolute change in weekly average of daily PP-NRS from parent study baseline | Parent study baseline to Week 48
  The PP-NRS is a validated single item 0-10 numeric rating scale assessing peak pruritus (itch) associated with AD with 0 = no itch and 10 = worst itch imaginable.
Non-responders from parent studies: Absolute change in weekly average of daily SD-NRS from parent study baseline | Parent study baseline to Week 48
  The SD-NRS is a single item 0-10 numeric rating scale assessing sleep disturbance associated with AD with 0 = no sleep loss and 10 = did not sleep at all.
Non-responders from parent studies: Proportion of participants with ≥3 points reduction in weekly average of daily SD-NRS from parent study baseline | Parent study baseline to Week 48
  The SD-NRS is a single item 0-10 numeric rating scale assessing sleep disturbance associated with AD with 0 = no sleep loss and 10 = did not sleep at all.
Non-responders from parent studies: Proportion of participants with ≥ 4 points reduction in weekly average of daily SP-NRS from parent study baseline [ | Parent study baseline to Week 48
  The SP-NRS is a single item 0-10 numeric rating scale assessing skin pain associated with AD with 0 = no pain and 10 = worst possible pain imaginable.
Non-responders from parent studies: Absolute change in weekly average of daily SP-NRS from parent study baseline | Parent study baseline to Week 48
  The SP-NRS is a single item 0-10 numeric rating scale assessing skin pain associated with AD with 0 = no pain and 10 = worst possible pain imaginable.
Non-responders from parent studies: Proportion of participants with a reduction in CDLQI ≥6^ among participants aged ≥12 to <16 years old and with CDLQI ≥6 at parent study baseline | Parent study baseline to Week 48
  The CDLQI is a validated 10-item questionnaire to measure dermatology-specific quality of life (QoL) in adult patients. Overall scoring ranges from 0 to 30, with a higher score indicating a poorer QoL. The symbol ^ represents "based on parent study baseline".
Non-responders from parent studies: Change in CDLQI^ in participants with age ≥12 to <16 years old | Parent study baseline to Week 48
  The CDLQI is a validated 10-item questionnaire to measure dermatology-specific quality of life (QoL) in adult patients. Overall scoring ranges from 0 to 30, with a higher score indicating a poorer QoL. The symbol ^ represents "based on parent study baseline".
Non-responders from parent studies: Change in DLQI^ in participants with age ≥16 years among the participants with DLQI ≥4 at parent study baseline | Parent study baseline to Week 48
  The DLQI is a validated 10-item questionnaire to measure dermatology-specific quality of life (QoL) in adult patients. Overall scoring ranges from 0 to 30, with a higher score indicating a poorer QoL. The symbol ^ represents "based on parent study baseline".
Non-responders from parent studies: Proportion of participants with ≥4 points reduction in DLQI from parent study baseline among the participants with DLQI ≥4 at parent study baseline | Parent study baseline to Week 48
  The DLQI is a validated 10-item questionnaire to measure dermatology-specific quality of life (QoL) in adult patients. Overall scoring ranges from 0 to 30, with a higher score indicating a poorer QoL.
Non-responders from parent studies: Proportion of participants with HADS-D <8 among the participants who had HADS-D ≥8 at parent study baseline | Parent study baseline to Week 48
  The Hospital Anxiety Depression Scale-Depression (HADS-D) ranges 0-21 with higher score indicating a poorer state.
Non-responders from parent studies: Proportion of participants with HADS-A <8 among the participants who had HADS-A ≥8 at parent study baseline | Parent study baseline to Week 48
  The Hospital Anxiety Depression Scale-Anxiety (HADS-A) ranges 0-21 with higher score indicating a poorer state.
All participants: Percentage of participants who experienced Treatment-Emergent Adverse Events (TEAEs), Treatment-Emergent Serious Adverse Events (TESAEs) and/or Treatment-Emergent Adverse Events of Special Interest (AESI) | Up to week 68
All participants: Serum amlitelimab concentrations measured at prespecified timepoints | Up to Week 68
All participants: Incidence of antidrug antibodies (ADAs) of amlitelimab | Up to Week 68

CONTACTS AND LOCATIONS:
Locations (326):
- United States (82):
  - Cahaba Dermatology & Skin Health Center- Site Number : 8401066, Birmingham, Alabama
  - Center for Dermatology and Plastic Surgery- Site Number : 8401119, Scottsdale, Arizona
  - Scottsdale Clinical Trials- Site Number : 8401149, Scottsdale, Arizona
  - Eclipse Clinical Research- Site Number : 8401158, Tucson, Arizona
  - Johnson Dermatology- Site Number : 8401076, Fort Smith, Arkansas
  - Encino Research Center- Site Number : 8401042, Encino, California
  - First OC Dermatology- Site Number : 8401025, Fountain Valley, California
  - Center for Dermatology Clinical Research- Site Number : 8401018, Fremont, California
  - Marvel Clinical Research- Site Number : 8401102, Huntington Beach, California
  - Sunwise Clinical Research- Site Number : 8401022, Lafayette, California
  - Torrance Clinical Research - Narbonne Avenue- Site Number : 8401027, Lomita, California
  - Dermatology Research Associates - Los Angeles- Site Number : 8401092, Los Angeles, California
  - LA Universal Research Center- Site Number : 8401064, Los Angeles, California
  - Northridge Clinical Trials - Northridge- Site Number : 8401080, Northridge, California
  - Cura Clinical Research - Oxnard- Site Number : 8401142, Oxnard, California
  - Southern California Dermatology- Site Number : 8401043, Santa Ana, California
  - Clinical Science Institute- Site Number : 8401028, Santa Monica, California
  - UConn Health - Farmington- Site Number : 8401115, Farmington, Connecticut
  - Pediatric Skin Research- Site Number : 8401198, Coral Gables, Florida
  - St. Jude Clinical Research- Site Number : 8401287, Doral, Florida
  - Beth Israel Deaconess Medical Center - Fort Myers- Site Number : 8401286, Fort Myers, Florida
  - Direct Helpers Research Center- Site Number : 8401056, Hialeah, Florida
  - Encore Medical Research - Hollywood- Site Number : 8401030, Hollywood, Florida
  - Clever Medical Research- Site Number : 8401160, Miami, Florida
  - Acevedo Clinical Research Associates- Site Number : 8401088, Miami, Florida
  - Florida International Research Center- Site Number : 8401091, Miami, Florida
  - Miami Dermatology and Laser Research - Miami - Southwest 87th Avenue- Site Number : 8401086, Miami, Florida
  - Anchor Medical Research- Site Number : 8401300, Miami, Florida
  - Savin Medical Group - Miami Lakes- Site Number : 8401085, Miami Lakes, Florida
  - Nuline Clinical Trial Center- Site Number : 8401161, Pompano Beach, Florida
  - Global Clinical Professionals (GCP)- Site Number : 8401045, St. Petersburg, Florida
  - Clinical Research Trials of Florida- Site Number : 8401023, Tampa, Florida
  - AllerVie Clinical Research - Columbus- Site Number : 8401104, Columbus, Georgia
  - Cleaver Medical Group- Site Number : 8401138, Dawsonville, Georgia
  - First Georgia Physician Group- Site Number : 8401190, Fayetteville, Georgia
  - Skin Care Physicians of Georgia - Macon- Site Number : 8401034, Macon, Georgia
  - Javara Research - Thomasville- Site Number : 8401189, Thomasville, Georgia
  - Rophe Adult & Pediatric Medicine- Site Number : 8401289, Union City, Georgia
  - NorthShore University Health System - Endeavor Health Medical Group - Skokie - Woods Drive- Site Number : 8401038, Skokie, Illinois
  - Dawes Fretzin Clinical Research- Site Number : 8401015, Indianapolis, Indiana
  - Equity Medical - Bowling Green- Site Number : 8401296, Bowling Green, Kentucky
  - Skin Sciences- Site Number : 8401039, Louisville, Kentucky
  - MedPharmics - Covington- Site Number : 8401137, Covington, Louisiana
  - BRCR Global Gretna- Site Number : 8401243, Gretna, Louisiana
  - Velocity Clinical Research - Lafayette- Site Number : 8401152, Lafayette, Louisiana
  - MetroBoston Clinical Partners - Brighton- Site Number : 8401128, Brighton, Massachusetts
  - Henry Ford Hospital- Site Number : 8401044, Detroit, Michigan
  - Revival Research Institute - Troy- Site Number : 8401012, Troy, Michigan
  - Oakland Medical Center- Site Number : 8401116, Troy, Michigan
  - Allergy & Immunology Associates of Ann Arbor- Site Number : 8401078, Ypsilanti, Michigan
  - SKY Integrative Medical Center/SKYCRNG - Ridgeland- Site Number : 8401058, Ridgeland, Mississippi
  - Skin Specialists- Site Number : 8401068, Omaha, Nebraska
  - Jubilee Clinical Research- Site Number : 8401054, Las Vegas, Nevada
  - Care Access - Hoboken- Site Number : 8401132, Hoboken, New Jersey
  - The University of New Mexico- Site Number : 8401263, Albuquerque, New Mexico
  - Equity Medical- Site Number : 8401239, New York, New York
  - Icahn School of Medicine at Mount Sinai- Site Number : 8401129, New York, New York
  - Sadick Research Group - New York - Park Avenue- Site Number : 8401050, New York, New York
  - OptiSkin- Site Number : 8401163, New York, New York
  - AXIS Clinicals - Fargo- Site Number : 8401196, Fargo, North Dakota
  - Bexley Dermatology Research- Site Number : 8401051, Bexley, Ohio
  - Apex Clinical Research Center- Site Number : 8401237, Mayfield Heights, Ohio
  - Oregon Medical Research Center- Site Number : 8401017, Portland, Oregon
  - Best Skin Research - Camp Hill- Site Number : 8401031, Camp Hill, Pennsylvania
  - Paddington Testing Company- Site Number : 8401041, Philadelphia, Pennsylvania
  - Clinical Research of Philadelphia- Site Number : 8401193, Philadelphia, Pennsylvania
  - Dermatology Associates of Plymouth Meeting- Site Number : 8401147, Plymouth Meeting, Pennsylvania
  - Columbia Dermatology & Aesthetics- Site Number : 8401166, Columbia, South Carolina
  - Tribe Clinical Research - Greenville - Verdae Boulevard- Site Number : 8401225, Greenville, South Carolina
  - Health Concepts- Site Number : 8401059, Rapid City, South Dakota
  - Arlington Research Center- Site Number : 8401248, Arlington, Texas
  - Dermatology Treatment and Research Center- Site Number : 8401164, Dallas, Texas
  - Derm Texas- Site Number : 8401217, Dallas, Texas
  - Prolato Clinical Research Center- Site Number : 8401209, Houston, Texas
  - SMS Clinical Research- Site Number : 8401182, Mesquite, Texas
  - Synapse Clinical Research - Missouri City- Site Number : 8401148, Missouri City, Texas
  - Texas Dermatology and Laser Specialists - San Antonio - Oakwell Court- Site Number : 8401131, San Antonio, Texas
  - Stryde Research - Epiphany Dermatology- Site Number : 8401185, Southlake, Texas
  - Complete Dermatology - Sugar Land- Site Number : 8401061, Sugar Land, Texas
  - Tanner Clinic - Layton Antelope A- Site Number : 8401151, Layton, Utah
  - Care Access - Arlington- Site Number : 8401134, Arlington, Virginia
  - Virginia Dermatology & Skin Cancer Center- Site Number : 8401047, Norfolk, Virginia
- Argentina (22):
  - Investigational Site Number : 0320021, Berazategui, Buenos Aires
  - Investigational Site Number : 0320017, Pilar, Buenos Aires
  - Investigational Site Number : 0320006, Rosario, Santa Fe Province
  - Investigational Site Number : 0320007, Rosario, Santa Fe Province
  - Investigational Site Number : 0320015, Rosario, Santa Fe Province
  - Investigational Site Number : 0320024, San Miguel de Tucumán, Tucumán Province
  - Investigational Site Number : 0320020, San Miguel de Tucumán, Tucumán Province
  - Investigational Site Number : 0320022, Buenos Aires
  - Investigational Site Number : 0320023, Buenos Aires
  - Investigational Site Number : 0320011, Buenos Aires
  - Investigational Site Number : 0320016, Buenos Aires
  - Investigational Site Number : 0320008, Buenos Aires
  - Investigational Site Number : 0320001, Buenos Aires
  - Investigational Site Number : 0320018, Buenos Aires
  - Investigational Site Number : 0320010, Buenos Aires
  - Investigational Site Number : 0320002, Buenos Aires
  - Investigational Site Number : 0320004, Buenos Aires
  - Investigational Site Number : 0320009, Buenos Aires
  - Investigational Site Number : 0320019, Buenos Aires
  - Investigational Site Number : 0320005, Buenos Aires
  - Investigational Site Number : 0320012, Corrientes
  - Investigational Site Number : 0320013, Mendoza
- Australia (5):
  - Investigational Site Number : 0360010, Westmead, New South Wales
  - Investigational Site Number : 0360007, Woolloongabba, Queensland
  - Investigational Site Number : 0360008, Melbourne, Victoria
  - Investigational Site Number : 0360006, Melbourne, Victoria
  - Investigational Site Number : 0361006, Traralgon, Victoria
- Brazil (14):
  - Centro de Diagnostico e Pesquisa da Osteoporose do Espirito Santo- Site Number : 0760017, Vitória, Espírito Santo
  - Centro de Pesquisas da Clínica IBIS- Site Number : 0760002, Salvador, Estado de Bahia
  - Hospital São Domingos- Site Number : 0760028, Bequimão, Maranhão
  - Hospital de Clinicas da Universidade Federal do Parana- Site Number : 0760022, Curitiba, Paraná
  - PUC Trials- Nucleo de Pesquisa clinica da Escola de Medicina da PUCPR- Site Number : 0760023, Curitiba, Paraná
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre- Site Number : 0760005, Porto Alegre, Rio Grande do Sul
  - Hospital São Lucas da PUCRS - Porto Alegre - Avenida Ipiranga- Site Number : 0760024, Porto Alegre, Rio Grande do Sul
  - Hospital das Clinicas da Faculdade de Medicina de Ribeirao Preto- Site Number : 0760015, Ribeirão Preto, São Paulo
  - Faculdade de Medicina do ABC- Site Number : 0760001, Santo André, São Paulo
  - Clinica de Alergia Martti Antila- Site Number : 0760006, Sorocaba, São Paulo
  - CCBR / IBPClin - Instituto Brasil de Pesquisa Clínica- Site Number : 0760018, Rio de Janeiro
  - Hospital Alemao Oswaldo Cruz - São Paulo- Site Number : 0760010, São Paulo
  - Centro de Desenvolvimento em Estudos ClÌnicos Brasil- Site Number : 0760014, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo- Site Number : 0760012, São Paulo
- Bulgaria (3):
  - Investigational Site Number : 1002007, Dupnitsa
  - Investigational Site Number : 1002004, Pleven
  - Investigational Site Number : 1002005, Sofia
- Canada (20):
  - Investigational Site Number : 1240039, Calgary, Alberta
  - Investigational Site Number : 1240031, Edmonton, Alberta
  - Investigational Site Number : 1240045, Red Deer, Alberta
  - Investigational Site Number : 1240046, Kelowna, British Columbia
  - Investigational Site Number : 1240040, Surrey, British Columbia
  - Investigational Site Number : 1240030, Surrey, British Columbia
  - Investigational Site Number : 1240041, Winnipeg, Manitoba
  - Investigational Site Number : 1240033, Ajax, Ontario
  - Investigational Site Number : 1240029, London, Ontario
  - Investigational Site Number : 1241106, Markham, Ontario
  - Investigational Site Number : 1240008, Mississauga, Ontario
  - Investigational Site Number : 1241108, Niagara Falls, Ontario
  - Investigational Site Number : 1240034, Ottawa, Ontario
  - Investigational Site Number : 1240038, Richmond Hill, Ontario
  - Investigational Site Number : 1240012, Toronto, Ontario
  - Investigational Site Number : 1240035, Toronto, Ontario
  - Investigational Site Number : 1241107, Waterloo, Ontario
  - Investigational Site Number : 1240006, Québec, Quebec
  - Investigational Site Number : 1240028, Regina, Saskatchewan
  - Investigational Site Number : 1240036, Saskatoon, Saskatchewan
- Chile (14):
  - Investigational Site Number : 1520004, Valdivia, Los Ríos Region
  - Investigational Site Number : 1520009, Osorno, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520013, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520008, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520002, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520003, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520014, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520010, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520011, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520005, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520001, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520015, Quillota, Región de Valparaíso
  - Investigational Site Number : 1520006, Viña del Mar, Región de Valparaíso
  - Investigational Site Number : 1520012, Talcahuano, Región del Biobío
- China (29):
  - Investigational Site Number : 1560042, Beijing
  - Investigational Site Number : 1560004, Beijing
  - Investigational Site Number : 1560030, Beijing
  - Investigational Site Number : 1560050, Changsha
  - Investigational Site Number : 1560022, Chengdu
  - Investigational Site Number : 1560060, Chengdu
  - Investigational Site Number : 1560068, Chengdu
  - Investigational Site Number : 1560057, Chongqing
  - Investigational Site Number : 1560065, Chongqing
  - Investigational Site Number : 1560043, Fuzhou
  - Investigational Site Number : 1560021, Guangzhou
  - Investigational Site Number : 1560025, Guangzhou
  - Investigational Site Number : 1560058, Guangzhou
  - Investigational Site Number : 1560044, Hangzhou
  - Investigational Site Number : 1560002, Hangzhou
  - Investigational Site Number : 1560006, Hangzhou
  - Investigational Site Number : 1560029, Hangzhou
  - Investigational Site Number : 1560007, Jinan
  - Investigational Site Number : 1560051, Nanchang
  - Investigational Site Number : 1560024, Ningbo
  - Investigational Site Number : 1560001, Shanghai
  - Investigational Site Number : 1560005, Shanghai
  - Investigational Site Number : 1560041, Shenyang
  - Investigational Site Number : 1560026, Shenyang
  - Investigational Site Number : 1560064, Shenzhen
  - Investigational Site Number : 1560023, Wenzhou
  - Investigational Site Number : 1560049, Wuhan
  - Investigational Site Number : 1560003, Wuxi
  - Investigational Site Number : 1560028, Zhenjiang
- Czechia (8):
  - Investigational Site Number : 2032106, Kutná Hora
  - Investigational Site Number : 2032105, Nový Jičín
  - Investigational Site Number : 2030010, Olomouc
  - Investigational Site Number : 2032104, Ostrava
  - Investigational Site Number : 2030009, Pilsen
  - Investigational Site Number : 2030008, Prague
  - Investigational Site Number : 2030011, Prague
  - Investigational Site Number : 2030006, Prague
- Denmark (3):
  - Investigational Site Number : 2080002, Aalborg
  - Investigational Site Number : 2080001, Aarhus
  - Investigational Site Number : 2080003, Herlev
- France (8):
  - Investigational Site Number : 2500008, Antony
  - Investigational Site Number : 2500013, Nice
  - Investigational Site Number : 2500003, Paris
  - Investigational Site Number : 2500006, Pierre-Bénite
  - Investigational Site Number : 2500007, Reims
  - Investigational Site Number : 2500010, Romans-sur-Isère
  - Investigational Site Number : 2500012, Rouen
  - Investigational Site Number : 2500002, Toulouse
- Germany (8):
  - Investigational Site Number : 2760020, Augsburg
  - Investigational Site Number : 2760009, Bad Bentheim
  - Investigational Site Number : 2760017, Hamburg
  - Investigational Site Number : 2760021, Hamburg
  - Investigational Site Number : 2762208, Kiel
  - Investigational Site Number : 2760016, Mainz
  - Investigational Site Number : 2762201, Münster
  - Investigational Site Number : 2760019, Witten
- Greece (2):
  - Investigational Site Number : 3000001, Athens
  - Investigational Site Number : 3000002, Thessaloniki
- India (7):
  - Investigational Site Number : 3560001, Ahmedabad
  - Investigational Site Number : 3560005, Belagavi
  - Investigational Site Number : 3560004, Chandigarh
  - Investigational Site Number : 3560006, Faridabad
  - Investigational Site Number : 3560007, Kolkata
  - Investigational Site Number : 3560002, Nagpur
  - Investigational Site Number : 3560003, Pune
- Israel (6):
  - Investigational Site Number : 3760004, Afula
  - Investigational Site Number : 3760005, Beersheba
  - Investigational Site Number : 3760001, Haifa
  - Investigational Site Number : 3760003, Jerusalem
  - Investigational Site Number : 3760006, Petah Tikva
  - Investigational Site Number : 3760002, Petah Tikva
- Italy (8):
  - Investigational Site Number : 3800003, Milan, Milano
  - Investigational Site Number : 3800018, Rozzano, Milano
  - Investigational Site Number : 3800013, Rome, Roma
  - Investigational Site Number : 3800012, Bologna
  - Investigational Site Number : 3800009, Catania
  - Investigational Site Number : 3800011, L’Aquila
  - Investigational Site Number : 3800008, Pisa
  - Investigational Site Number : 3800022, Vicenza
- Japan (18):
  - Investigational Site Number : 3920009, Chitose, Hokkaido
  - Investigational Site Number : 3923114, Obihiro, Hokkaido
  - Investigational Site Number : 3920008, Sapporo, Hokkaido
  - Investigational Site Number : 3920006, Kobe, Hyōgo
  - Investigational Site Number : 3920005, Sagamihara, Kanagawa
  - Investigational Site Number : 3923113, Yokohama, Kanagawa
  - Investigational Site Number : 3920010, Miyagi-gun, Miyagi
  - Investigational Site Number : 3920011, Sendai, Miyagi
  - Investigational Site Number : 3923109, Habikino, Osaka
  - Investigational Site Number : 3923110, Sakai, Osaka
  - Investigational Site Number : 3920002, Iruma, Saitama
  - Investigational Site Number : 3923106, Mibu, Tochigi
  - Investigational Site Number : 3920004, Chūō, Tokyo
  - Investigational Site Number : 3923107, Minato, Tokyo
  - Investigational Site Number : 3920001, Tachikawa, Tokyo
  - Investigational Site Number : 3923108, Kagoshima
  - Investigational Site Number : 3923102, Kyoto
  - Investigational Site Number : 3920003, Kyoto
- Mexico (5):
  - Investigational Site Number : 4840011, Monterrey, Nuevo León
  - Investigational Site Number : 4840005, Monterrey, Nuevo León
  - Investigational Site Number : 4840012, Aguascalientes
  - Investigational Site Number : 4840009, Durango
  - Investigational Site Number : 4840003, Veracruz
- Poland (8):
  - Investigational Site Number : 6162406, Krakow, Lesser Poland Voivodeship
  - Investigational Site Number : 6160010, Tarnów, Lesser Poland Voivodeship
  - Investigational Site Number : 6160004, Lublin, Lublin Voivodeship
  - Investigational Site Number : 6160002, Lodz, Lódzkie
  - Investigational Site Number : 6160009, Warsaw, Masovian Voivodeship
  - Investigational Site Number : 6160007, Warsaw, Masovian Voivodeship
  - Investigational Site Number : 6160006, Gdansk, Pomeranian Voivodeship
  - Investigational Site Number : 6160003, Katowice, Silesian Voivodeship
- Portugal (4):
  - Investigational Site Number : 6200005, Lisbon
  - Investigational Site Number : 6200004, Lisbon
  - Investigational Site Number : 6200001, Lisbon
  - Investigational Site Number : 6200003, Porto
- South Africa (7):
  - Investigational Site Number : 7100015, Benoni
  - Investigational Site Number : 7100010, Cape Town
  - Investigational Site Number : 7100009, Cape Town
  - Investigational Site Number : 7100012, Durban
  - Investigational Site Number : 7100001, Durban
  - Investigational Site Number : 7100007, Johannesburg
  - Investigational Site Number : 7100003, Pretoria
- South Korea (13):
  - Investigational Site Number : 4100008, Daegu, Daegu
  - Investigational Site Number : 4100012, Gwangju, Gwangju
  - Investigational Site Number : 4100002, Ansan-si, Gyeonggi-do
  - Investigational Site Number : 4100014, Seongnam-si, Gyeonggi-do
  - Investigational Site Number : 4100009, Suwon, Gyeonggi-do
  - Investigational Site Number : 4100003, Yangsan, Gyeongsangnam-do
  - Investigational Site Number : 4100015, Bupyeong-gu, Incheon-gwangyeoksi
  - Investigational Site Number : 4100010, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100013, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100007, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100006, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100011, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100017, Seoul, Seoul-teukbyeolsi
- Spain (12):
  - Investigational Site Number : 7240010, Esplugues de Llobregat, Barcelona [Barcelona]
  - Investigational Site Number : 7240008, Bilbao, Basque Country
  - Investigational Site Number : 7240012, Las Palmas de Gran Canaria, Las Palmas
  - Investigational Site Number : 7240015, Pamplona, Navarre
  - Investigational Site Number : 7240014, Vigo, Pontevedra [Pontevedra]
  - Investigational Site Number : 7240020, Seville, Sevilla
  - Investigational Site Number : 7240023, Burjassot - Valencia, Valenciana, Comunidad
  - Investigational Site Number : 7242505, Alicante
  - Investigational Site Number : 7240018, Granada
  - Investigational Site Number : 7240019, Granada
  - Investigational Site Number : 7240029, Madrid
  - Investigational Site Number : 7242503, Madrid
- Sweden (2):
  - Investigational Site Number : 7520006, Älvsjö
  - Investigational Site Number : 7520001, Örebro
- Taiwan (4):
  - Investigational Site Number : 1583201, Kaohsiung City
  - Investigational Site Number : 1583202, Taichung
  - Investigational Site Number : 1580001, Taipei
  - Investigational Site Number : 1580003, Taipei
- Turkey (Türkiye) (9):
  - Investigational Site Number : 7920001, Antalya
  - Investigational Site Number : 7920008, Gaziantep
  - Investigational Site Number : 7920005, Istanbul
  - Investigational Site Number : 7920006, Istanbul
  - Investigational Site Number : 7920002, Istanbul
  - Investigational Site Number : 7920009, Istanbul
  - Investigational Site Number : 7920004, Kayseri
  - Investigational Site Number : 7920011, Mersin
  - Investigational Site Number : 7920007, Samsun
- United Kingdom (5):
  - Investigational Site Number : 8260003, Portsmouth, Hampshire
  - Investigational Site Number : 8260004, Leicester, Leicestershire
  - Investigational Site Number : 8262601, London, London, City of
  - Investigational Site Number : 8262602, London, London, City of
  - Investigational Site Number : 8260006, Glasgow

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: EFC17600 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25741&tenant=MT_SNY_9011